CLINICAL TRIAL: NCT05260086
Title: Untersuchung Von Hirnnetzwerken Durch Nicht-invasive Transkranielle Magnetstimulation - Phase 2 (PreNeSt2)
Brief Title: Pre-mapping Networks for Brain Stimulation 2
Acronym: PreNeSt2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, PD Dr. Roberto Goya-Maldonado, Principal Investigator, University Medical Center Goettingen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01759
Record Dates: First submitted 2021-12-10; First posted 2022-03-02 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Depressive Episode; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The investigators compare study outcomes using aiTBS in personalized stimulation targets vs conventional F3 stimulation targets in parallel arms, each arm controlled by its respective sham stimulation in a counterbalanced crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized aiTBS active - sham (Experimental): counterbalanced crossover with sham neuronavigated stimulation
  Interventions: Device: Neuronavigated aiTBS
- Conventional (F3) aiTBS active - sham (Active Comparator): counterbalanced crossover with sham neuronavigated stimulation
  Interventions: Device: Neuronavigated aiTBS

INTERVENTIONS:
Device: Neuronavigated aiTBS — Accelerated intermittent theta burst stimulation (aiTBS, 4 sessions per day with at least 20 minutes pause between sessions) in the left dorsolateral prefrontal cortex (DLPFC)

SUMMARY:
The investigators compare the primary and secondary outcome measures using accelerated intermittent theta burst stimulation (aiTBS, 20 sessions active and 20 sessions sham in a counterbalanced crossover design) to treat depressive symptoms with 2 parallel arms of intervention: personalized (stimulation position based on participants' brain networks) vs conventional (stimulation in F3 position of the 10-20 EEG cap) aiTBS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 60 years
* Diagnosis of major depressive disorder according to DSM 5 (F32.x according to ICD-10) or bipolar disorder (bipolar I or bipolar II) according to DSM 5 (F31.x according to ICD-10) and an acute depressive condition at the time of the initial examination in outpatient or inpatient treatment (e.g. Department of Psychiatry and Psychotherapy, UMG)
* Availability of informed consent to participate in the study, including the examinations and interventions

Exclusion Criteria:

* Neurological diseases, current or previous
* Other Axis I diagnoses that mimic the affective disorder, current or previous
* Physical illnesses that could be related to the affective symptoms (so-called organic causes)
* Illicit drug use in the past month
* Substance dependence, current or previous
* Physical illnesses which, depending on their type and severity, could interfere with the planned examinations, influence the parameters to be examined or endanger the test participant during the course of the examination
* Medical contraindications against performing an MRT examination / rTMS application (such as metal parts in the body, e.g. implants, pacemakers, infusion pumps, metal splinters, etc.)
* Pregnancy
* Previously known cerebral-morphological abnormalities (e.g. tumor, lesion, etc.)
* Evidence or history of epilepsy
* Head trauma with a history of loss of consciousness
* Unwillingness to be informed of incidental findings
* Participation in an rTMS / EKT application within the last 8 weeks
* Lack of the ability to provide informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS scores in units of scale) | 6 weeks
  Administer Rating Scale
heart rate and its variability in RR slope and RMSSD values | 4-6 weeks
  Potential marker of treatment response

SECONDARY OUTCOMES:
Hamilton Rating Scale for Depression (HAMD-17 scores in units of scale) | 6 weeks
  Administer Rating Scale
Beck Depression Inventory (BDI-2 scores in units of scale) | 6 weeks
  Self Rating Scale
DMN decoupling / other networks in rho and z values | 4-6 weeks
  Potential markers of treatment response
epi / genetic markers of neuroplasticity in ng | 5-6 weeks
  Potential markers of treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Goya-Maldonado, MD, Principal Investigator — University Medical Center Göttingen (UMG)
Locations (1):
- Laboratory of Systems Neuroscience and Imaging in Psychiatry (SNIP-Lab Göttingen), Göttingen, Germany